CLINICAL TRIAL: NCT06974513
Title: Auditory Localization in Virtual Reality in Patients With a First Episode of Psychosis
Brief Title: Auditory Localization in Schizophrenia
Acronym: LOCIZ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A00469-40; PRVR06 (Other Grant/Funding Number: Centre Hospitalier le Vinatier)
Record Dates: First submitted 2025-04-29; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Auditory Perception
Keywords: Localization; Auditory perception; Source monitoring; Virtual reality

STUDY DESIGN:
Intervention Model Description: 30 patients with a first episode psychosis and 30 healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group with a first episode psychosis (Experimental): Tasks will include an auditory localization task performed in virtual reality, a source-monitoring task, an externalization task and a battery of psychoacoustic tests.
  Interventions: Behavioral: cognitive experiments' session
- Healthy control subjects (Active Comparator): Tasks will include an auditory localization task performed in virtual reality, a source-monitoring task, an externalization task and a battery of psychoacoustic tests.
  Interventions: Behavioral: cognitive experiments' session

INTERVENTIONS:
Behavioral: cognitive experiments' session — The aim of this unique session of cognitive experiments is to study the auditory localization performance in patients with a first episode of psychosis. Results of this Arm 1 will be compared to those of Arm 2.

SUMMARY:
Auditory sound localization is the ability to identify the position of a sound source in space. It is defined into 3 dimensions: by its position in azimuth, elevation and distance. If it is difficult to localize a sound source, it is possible to remove the localization ambiguity by interacting with the environment, in particular by changing one's position in relation to the source (e.g. by changing the orientation of the head).

Patients with schizophrenia have difficulties to localize and discriminate sounds in space but it is still poorly explored.

Additionally, deficits in auditory localization could underlie difficulties in source-monitoring (i.e., distinguish the source/origin of the information) reported in schizophrenia or deficits in auditory externalization (i.e., perception of sound outside the head).

Furthermore, schizophrenia is characterized by cerebral abnormalities in the auditory cortex, manifesting as auditory processing disorders at different stages of the pathology. Auditory localization may therefore be impaired from the onset of a first psychotic episode (FEP). This early phase of the disease is also referred to as the "critical" period, as the chances of remission are highest and the response to treatment is best. However, the three-dimensional aspect of auditory perception and the behavioral exploration strategies used to localize a sound in the early stages of schizophrenia are still little studied.

DETAILED DESCRIPTION:
The main objective of this study is to study the auditory localization performance on the horizontal and vertical planes (sound direction) in patients with a first episode psychosis (FEP) compared to healthy control subjects.

This study will:

* evaluate the role of head movement on auditory localization abilities in patients with FEP compared with healthy control subjects;
* evaluate the localization abilities of sounds in a noisy environment in patients with FEP compared with healthy control subjects;
* evaluate the repercussions of poor auditory localization performance on the ability to distinguish between what comes from an internal source and what comes from an external source (source-monitoring abilities);
* evaluate the repercussions of poor auditory localization performance on the ability to externalize an external auditory source compared with an internal source (auditory externalization abilities);
* evaluate the relationships between auditory localization performance and auditory discrimination performance (pitch, volume, length);
* evaluate the repercussions of the severity of symptoms in patients with FEP on auditory localization performance.

Subjects will undergo several auditory and cognitive tasks. The duration of the entire experiments will be 2.30 hours:

* An auditory localization task in virtual reality with the SPHERE paradigm: the subject is immerged into a room and sounds are delivered through loudspeakers in different localization on the horizontal and vertical planes. Sounds are delivered in two experimental blocks: silent and noisy background. Each block is divided into two listening conditions: fixed head and active head movement (i.e., with the possibility of moving the head). Subjects have to localize each sound.
* A source monitoring task divided into two parts: one part that will evaluate the reality-monitoring performances ('hear-imagine' task). Subjects either have to listen to words or imagine themselves listening to words; Another part evaluating internal source-monitoring performances ('say-imagine' task). Subjects either have to pronounce words or imagine themselves pronouncing words.
* An auditory externalization task: Nonverbal sounds are delivered through headphones and processed to be perceived inside or outside the head. Subjects will have to discern whether a sound is perceived as coming from inside or outside the head.
* A battery of psychoacoustic tests including the Tone Matching Task (TMT) which evaluates the capacity of discriminating static pitch.

ELIGIBILITY:
Inclusion Criteria:

* Informed of the study and having signed the consent form
* With normal vision (with or without correction)
* Able to understand the experimental instructions
* Affiliated to the social security system
* French language spoken, read and written

Exclusion Criteria:

* Patients with a DSM-5 diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder or brief psychotic disorder
* Early intervention for first psychotic episodes

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Auditory localization performance in virtual reality | Baseline
  an auditory localization task in virtual reality was design for this study. Sounds are presented in different localization on the horizontal and vertical planes. Participants performed two blocks (noise, silent background) divided into two conditions (localization with the fixed head or with the possibility of moving the head). Participants have to determine the localization of sound in space. The main outcome will be the perception performance corresponding to the directionality error (2Dd error in cm) in relation to the sound source.

SECONDARY OUTCOMES:
The impact of head movements on auditory localization performance | Baseline
  an auditory localization task in virtual reality was design for this study. Participants have to determine the localization of sounds in two different conditions: fixed head or with the possibility of moving the head. The main outcome will be the perception performance corresponding to the directionality error (2Dd error in cm) in the two different conditions.
The impact of background noise on auditory localization performance | Baseline
  an auditory localization task in virtual reality was design for this study. Participants have to determine the localization of sounds in two different blocks: silent and noisy background. The main outcome will be the perception performance corresponding to the directionality error (2Dd error in cm) in the two different blocks.
Source-monitoring performance | Baseline
  A computerized source memory task was designed for this study to assess the reality-monitoring (distinguishing real source and imagined source) and et internal source-monitoring (distinguishing two internal sources). The rate of correct responses and inversions are the outcome.
Performance on auditory externalization | Baseline
  computerized auditory externalization task. Nonverbal sounds are presented, the azimuth is varied in order to create the impression of the sound coming either from inside or outside the head. Subjects have to determine whether the nonverbal burst was perceived as coming from inside or outside their head. The rate of correct responses (inside/outside) is the outcome.
Performance on basic auditory tasks | Baseline
  a computerized psychoacoustic battery of tests : Tone Matching Task (evaluating nonverbal pitch). The rate of correct responses is the outcome.
Performance on basic auditory tasks | Baseline
  a computerized psychoacoustic battery of tests : psychoacoustic tasks measuring amplitude. The rate of correct responses is the outcome.
Performance on basic auditory tasks | Baseline
  a computerized psychoacoustic battery of tests : psychoacoustic tasks measuring length of sound . The rate of correct responses is the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric HAESEBAERT, university professor, Principal Investigator — hopital le Vinatier
Locations (1):
- Centre hospitalier le Vinatier, Bron, France